CLINICAL TRIAL: NCT02465281
Title: Correlation Analysis Between Brain Lesions and Sensorimotor Impairments in Individuals With Stroke (Preliminary Study)
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1503M66381
Record Dates: First submitted 2015-05-29; First posted 2015-06-08 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Stroke patients: 20 patients who are at least 6 months post stroke. Device: 3T scanner with MRI-compatible robot
  Interventions: Other: Device: 3T scanner with MRI-compatible robot
- Healthy volunteers: 80 age-matched healthy volunteers
  Interventions: Other: Device: 3T scanner with MRI-compatible robot

INTERVENTIONS:
Other: Device: 3T scanner with MRI-compatible robot

SUMMARY:
The objective of the preliminary study is:

1. To identify correlations between brain lesions and sensorimotor impairments in stroke.
2. To identify possible patterns between brain lesions and sensorimotor impairments that might increase our understanding in stroke recovery and guide further tailor-based neuro-rehabilitation

DETAILED DESCRIPTION:
The purpose of this study is to investigate arm and hand function after stroke and how the location of the brain lesion affects arm and hand function. We are hoping to collect data in the form of assessments what you feel and how your arm moves, surveys about activities in daily life and well-being, and we will perform 1 Magnetic Resonance Imaging (MRI) scan. MRI scans are loud but painless; nothing is injected. With MRI, we collect images from the brain.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for healthy subjects are:

  * medically stable;
  * 18 - 99 years of age;
  * able to hear the instructions given during the study

Inclusion criteria for stroke patients are:

* at least 6 months post-stroke;
* medically stable;
* 18 - 99 years of age;
* subcortical or cortical infarct confirmed with MRI;
* Mini-mental State Exam > 24/30 (Folstein et al., 1975);
* able to hear the instructions given during the study;
* able to comprehend the instructions given during the study;
* able to commit time to participate in a 6-12-weeks rehabilitation program

Exclusion Criteria:

Exclusion criteria for healthy subjects are:

* having ever experienced a stroke or another brain injury or illness related to the brain that has lasting effects or effects experienced at the moment of recruitment;
* severe sensory impairments such that different movements of the finger, hand or wrist are not reliably felt;
* contractures in tested arm that hinder persons from keeping the outstretched arm in a relaxed position;
* interfering comorbidities (e.g. fracture, cancer, peripheral neuropathy);
* exhibit contra-indications to enter the magnetic field of the 3T (pacemakers, metal parts in the body etc);
* pregnant or nursing mother;
* adults lacking capacity to consent

Exclusion criteria for stroke patients are:

* insular or cerebellar infarcts/brain lesions;
* unilateral spatial neglect, identified by a standard neuropsychological assessment (Bell's test (score/35, Gauthier et al., 1989);
* aphasia;
* apraxia (TULIA, Vanbellingen et al., 2011);
* severe sensory impairments such that different movements of the finger, hand or wrist are not reliably felt;
* contractures in the hemiplegic arm that hinder patients from keeping the outstretched arm in a relaxed position;
* interfering comorbidities (e.g. fracture, cancer, peripheral neuropathy);
* patients currently receiving therapy for their hemiplegic arm, the latter in order to avoid confounding treatment effects;
* exhibit contra-indications to enter the magnetic field of the 3T (pacemakers, metal parts in the body etc);
* pregnant or nursing mother;
* adults lacking capacity to consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Control Group Stroke patient subjects
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-09-23 (Actual); Study Completion 2016-09-23 (Actual)

PRIMARY OUTCOMES:
Structural and Functional Imaging | 1 week
  Identify correlations between brain lesions and sensimotor impairments in stroke
Identify Possible Patterns | 1 week
  Identify possible patterns between brain lesions and senosrimotor impairments that might increase our understanding in stroke recovery and guide further tailor-based neuro-rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Anne Van de Winckel, PhD, MS, PT, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States